CLINICAL TRIAL: NCT02109471
Title: Observational Study of Corneal Opacities in Adults
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, David Huang, David Huang, MD, PhD, Professor of Ophthalmology, Oregon Health and Science University, Oregon Health and Science University
Other Study IDs: OHSU IRB#6612 - Opac; R01EY018184 (NIH)
Record Dates: First submitted 2014-01-14; First posted 2014-04-10 (Estimated); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Corneal Opacities (Scar and Stromal Dystrophy)
Keywords: corneal opacities; Optical coherence tomography
MeSH Terms: conditions — Corneal Opacity; Cicatrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- corneal opacities

SUMMARY:
A prospective observational study on corneal opacities (scar and stromal dystrophy) in adults (n=150) will be conducted at OHSU. The Optovue anterior segment OCT will be used to perform 3-D corneal scans. These scans will be used to assess opacity depth and measure corneal thickness (pachymetry), corneal topography (anterior and posterior), and epithelial thickness maps. The ultrahigh-speed MIT OCT prototypes will also be used when they become available. A comprehensive eye examination, Placido-ring corneal topography, ultrasound pachymetry, and Scheimpflug camera imaging, will be performed for comparison.

ELIGIBILITY:
Inclusion Criteria:

• Adult (18 & older) patients presenting in OHSU Casey Eye Clinic with corneal opacities (scar and stromal dystrophy)

Exclusion Criteria:

* Inability to give informed consent.
* Inability to maintain stable fixation for OCT imaging.
* Inability to commit to required visits to complete the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting in OHSU Casey Eye Clinic with corneal opacities (scar and stromal dystrophy)
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identification of suitable subjects | 2 years
  The primary goal of this observational study is to identify suitable subjects for the clinical trials of OCT-guided transepithelial PTK.

SECONDARY OUTCOMES:
Validate OCT topography | 2 years
  A second goal is to validate OCT anterior topography by comparison with standard Placido-ring corneal topography and develop a mathematical model that relates epithelial thickness variation to corneal mean curvature.

CONTACTS AND LOCATIONS:
Overall Officials: David Huang, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Humberto Martinez, Portland, Oregon, United States